CLINICAL TRIAL: NCT00013637
Title: Lead Exposure, Genetics, and Osteoporosis Epidemiology
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8074-CP-001
Record Dates: First submitted 2001-03-26; First posted 2001-03-28 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Lead
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This study's primary objective is to assess the effects of environmental lead exposures and genetic risk factors on the development of osteoporosis in middle-aged women.

ELIGIBILITY:
Healthy participants in the Nurses' Health Study who live in the greater Boston metropolitan area.

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650
Dates: Start 1998-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States